CLINICAL TRIAL: NCT07393204
Title: Italian Real-world Study on Epcoritamab in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Italian Real-World Study of Epcoritamab in Relapsed or Refractory DLBCL
Acronym: EPKEY_HSR
Status: Active, not recruiting | Type: Observational
Sponsor: Andrés José Maria Ferreri (Other)
Responsible Party: Sponsor-Investigator, Andrés José Maria Ferreri, Director of Lymphoma Unit, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: EPKEY_HSR
Record Dates: First submitted 2025-12-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Relapsed Diffuse Large B-cell Lymphoma (DLBCL); Refractory Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; relapsed; refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epcoritamab treatment: Patients registered in the Cnn program of epcoritamab (between February 19, 2024 and September 25, 2024) that received at least 1 dose of this antibody.

SUMMARY:
This study describes the effectiveness of epcoritamab outside the clinical trial setting in pts with DLBCL relapsed or refractory after 2 or more previous lines of therapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients registered in the Cnn program of epcoritamab (between February 19, 2024 and September 25, 2024)
* Received at least one dose of epcoritamab
* Free and voluntary written informed consent

Exclusion Criteria:

* Age < 18 years
* Patients who received epcoritamab outside the Cnn program (e.g., open access program, compassionate use, off-label, prospective trials).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is expected to include approximately 150 patients. Patients registered in the Cnn program of epcoritamab (between February 19, 2024 and September 25, 2024) that received at least 1 dose of this antibody.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Response Rate (ORR), defined as the best objective response achieved during or after treatment with epcoritamab, according to Lugano Criteria

SECONDARY OUTCOMES:
Adverse Event according to CTCAE v5.0 | through study completion, an average of 1 year
  rate and severity of AEs (Adverse Event), AESIs (adverse events of special interest) and SAEs (Serious Adverse Event) according to the Common Terminology Criteria for Adverse Events (CTCAE v.5.0)
Incidence and Severity of Cytokine Release Syndrome (CRS) | through study completion, an average of 1 year
  Incidence and Severity of Cytokine Release Syndrome (CRS) according to ASTCT CRS grading criteria
Incidence and Severity of Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) | through study completion, an average of 1 year
  ICANS graded according to ASTCT ICANS grading criteria (ICE score)
Complete Response rate | through study completion, an average of 1 year
  CR rate defined as the proportion of patients with CR, according to Lugano Criteria at 1, 2, 3, 6, 9 and 12 months since treatment start
Duration of Response | through study completion, an average of 1 year
  DoR is defined as the time from the first documentation of response (CR or PR) to the date of PD or death, whichever occurs earlier.
Duration of Complete Response | through study completion, an average of 1 year
  DoCR is defined as the time from the first documentation of CR to the date of PD or death, whichever occurs earlier.
Progression Free Survival | through study completion, an average of 1 year
  PFS is defined as the time from the start of the treatment to first documented PD or death due to any cause, whichever occurs earlier.
Overall Survival | through study completion, an average of 1 year
  OS is defined as the time from the start of epcoritamab treatment to death
Time To Next Treatment | through study completion, an average of 1 year
  TTNT is defined as duration from treatment initiation to the start of new anti-lymphoma therapy or death due to PD, whichever occurs earlier
Duration of Treatment | through study completion, an average of 1 year
  Duration of Treatment (DoT) is defined as the time from the start of the treatment to discontinuation or death due to any cause, whichever occurs earlier.
Health Care Resource Utilization (HCRU) | through study completion, an average of 1 year
  Health Care Resource Utilization (HCRU) as number and duration of unplanned hospitalizations during treatment and follow-up, number of hematological visits, load of diagnostic exams

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided